CLINICAL TRIAL: NCT06209073
Title: Efficacy of Virtual Reality Exercises on Sarcopenia in Patients With Liver Transplantation
Acronym: LT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nabil Mahmoud Ismail Abdel-Aal, Principal Investigator: nabil mahmoud ismail abdel-Aal, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003915
Record Dates: First submitted 2023-12-28; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-01

CONDITIONS: Sarcopenia
Keywords: liver transplantation; virtual reality; quality of life
MeSH Terms: conditions — Sarcopenia | interventions — Exergaming

STUDY DESIGN:
Intervention Model Description: virtual reality and conventional treatment
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelop
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality exercise (Experimental): the patients will receive virtual reality and conventional therapy three times a week for six weeks
  Interventions: Other: Virtual Reality exercise; Other: conventional treatment
- conventional treatment (Experimental): the patients will receive conventional treatment three times a week for six weeks
  Interventions: Other: conventional treatment

INTERVENTIONS:
Other: Virtual Reality exercise — after explaining the treatment method for patients, the patients will perform full body aerobic exercise by applying kick boxing to destroy walls of rock; the patient moves most of body muscles in this game. He or she flex and extend the shoulder and the elbow with flexion and extension in the knee. squatting exercise, endurance exercise, coordination for arm and shoulder exercise will also performed in virtual reality
  Arms: virtual reality exercise
Other: conventional treatment — the patients will receive conventional treatment in the form of aerobic exercise, resistance exercise and endurance exercise.

SUMMARY:
This study will be conducted to investigate the effect of virtual reality exercises on hand grip strength, pinch strength, quadriceps muscle strength, exercise capacity, fatigue, and quality of life in patients with liver transplantation.

DETAILED DESCRIPTION:
Liver transplantation (LT) continues to prove to be the best choice for curing patients with end-stage liver disease (ESLD) . Management strategies in peri-transplantation care have significantly improved the outcomes of patients after LT. One of the most challenging tasks of LT is defining which patients are clinically appropriate for this therapy. Evaluating disease severity for patients with ESLD is a serious challenge for liver transplant surgeons, and there is a critical need for better methods of risk stratification. The most common complications involved include ascites, hepatic encephalopathy, and variceal bleeding; however, severe muscle wasting or sarcopenia is the most common and frequently undiagnosed complications that negatively impact survival, quality of life, and response to stressors, such as infections and surgeries. Virtual reality (VR) is an interactive, 3-dimensional computer experience occurring in real time. It allows the users to participate in multisensory and multidimensional virtual environments . It provides the participants with real-time auditory, visual, and proprioception sensory feedback. It also provides a safe virtual exercise environment. sixty patients with liver transplantation will be assigned randomly to two groups; experimental group will receive virtual reality exercise plus traditional therapy for six weeks, control group will receive traditional therapy alone for six weeks

ELIGIBILITY:
Inclusion Criteria:

Sixty patients suffer from sarcopenia with liver transplantation. The age of patients ranges from (18:65) years. All patients must be conscious. Patients suffer from muscle weakness Patients suffer from fatigue Patients with low muscle endurance Patients' cases must be stable to deal with them

Exclusion Criteria:

Patients will be excluded if they have any of the following:

Any sign of acute rejection of the transplanted organ Acute hemorrhage Electrolyte imbalance Physiological instability Sever neurologic complication Sever cardiovascular co-morbidities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-25 (Estimated); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Hand grip strength | up to six weeks
  JAMAR hand grip dynamometer will be used to measure hand grip strength

SECONDARY OUTCOMES:
Pinch strength | up to six weeks
  JAMAR Pinch grip dynamometer will be used to measure pinch strength
Respiratory function | up to six weeks
  spirometry will be used to measure the the ratio of forced expiratory volume in one second (FEV1) to forced vital capacity (FVC)
Fatigue | up to six weeks
  Arabic version of fatigue severity scale will be used to measure fatigue. It consists of 9 items , patients score each item from 1 to 7, based on the extent, to which they agree or disagree with each statement (1 = strong disagreement, 7 = strong agreement). The FSS can be scored either by obtaining a total score, or by calculating a mean score across all 9 items, with higher scores indicating more severe fatigue.
life disability | up to six weeks
  The World Health Organization Quality of Life - BREF (WHOQOL-BREF) will be used to assess quality of life.The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale.
exercise capacity | up to six weeks
  six minute walk test will be used to assess the exercise capacity.The 6-minute walk test requires a subject to walk as far as he or she can in 6 minutes, with rests as needed.
quadriceps strength | up to six weeks
  hand-held dynamometer (HHD) ( Lafayette Instrument Company, USA) will be used to assess quadriceps strength. it is a reliable strength testing equipment. It is a portable device that can be used to obtain more discrete, objective measures of strength during manual muscle testing

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Elshrief, Bsc, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt